CLINICAL TRIAL: NCT04646681
Title: Development of a Targeted Patient Portal Intervention to Improve Depression Treatment Adherence, Satisfaction, and Outcomes
Brief Title: Development of a Targeted Patient Portal Intervention to Improve Depression Treatment Adherence and Outcomes
Acronym: Patient Portal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolyn L Turvey (Other)
Responsible Party: Sponsor-Investigator, Carolyn L Turvey, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201805861
Record Dates: First submitted 2020-11-20; First posted 2020-11-30 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Depression
Keywords: patient portals; treatment adherence
MeSH Terms: conditions — Depression; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Behavioral: ConnectCare
- Group 2 (No Intervention)

INTERVENTIONS:
Behavioral: ConnectCare — increased monitoring between clinical mental health visits
  Arms: Group 1

SUMMARY:
The purpose of this research study is to learn how best to use patient portals to help improve the treatment of mood disorders.

DETAILED DESCRIPTION:
This study is being done in 3 phases. First 2 phases were observational with total enrollment of 300 subjects. The final 3rd phase is interventional and we are anticipating to enroll 50 subjects. It is described below.

Patients being treated for depressive symptoms at the University of Iowa, Department of Psychiatry are invited to participate. Participants will complete a remote (phone or video) visit. After being informed about the study and potential risks, those who consent to being in the study will be assigned to one of two groups. They will complete an online survey and receive some basic training on patient portals. After the visit. both groups will be followed for 6 months. Depending on their group assignment, they will complete:

* two to five phone calls with a study team member and
* two to five online questionnaires

ELIGIBILITY:
Inclusion Criteria:

* English speaking,
* PHQ-9 score of 10 or higher (questions 1-8 only),
* Taking medication for depressive symptoms,
* 1 or more appointments scheduled or planned with University of Iowa psychiatry provider in next 6 months,
* Home computer w/internet access,
* MyChart (University of Iowa Healthcare's patient portal) account/MyChart enrollment

Exclusion Criteria:

* Psychotic disorder/symptoms,
* Current substance use disorders (other than alcohol, tobacco, marijuana),
* Active suicidal ideation within past 1 year,
* Cognitive impairment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Once per month for 6 months
  measures the severity of depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Turvey, phD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Carver College of Medicine, Dept. of Psychiatry, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No